CLINICAL TRIAL: NCT00207090
Title: Effect of Rifampin on the Pharmacokinetics of Ixabepilone in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA163-102
Record Dates: First submitted 2005-09-12; First posted 2005-09-21 (Estimated); Results first posted 2010-10-01 (Estimated); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Advanced Solid Tumors; Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — ixabepilone; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ixabepilone + rifampin (Experimental)
  Interventions: Drug: ixabepilone; Drug: Rifampin

INTERVENTIONS:
Drug: ixabepilone — ixabepilone solution, intravenous, 40 mg/m2, once every 3 weeks until disease progression
  Other Names: IXEMPRA®; BMS-247550
Drug: Rifampin — rifampin tablets, oral, 600 mg once daily, only on Days 15 to 21 of Cycle 1 and Days 1 to 7 of Cycle 2

SUMMARY:
The purpose of this study is to test how rifampin affects the removal of BMS-247550 (ixabepilone) from the body.

ELIGIBILITY:
Inclusion Criteria:

* Up to three prior chemotherapy regimens
* Measurable or non-measurable disease
* Available for treatment and follow-up

Exclusion Criteria:

* Neuropathy
* Uncontrolled cardiovascular disease
* Refusal to participate in genetic analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2005-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 19 participants were enrolled and 15 were treated with the study drug. 4 participants were not treated (1 participant due to an adverse event [AE] and 3 participants for no longer meeting study criteria)
Groups:
- All Participants: All treated participants who received at least 1 dose of study drug. On Day 1 of Cycle 1, each participant received a single 3-hour IV infusion of ixabepilone 40 mg/m^2. On Day 15, participants were administered an oral dose of 600 mg rifampin in the clinic and on Days 16-21, participants self-administered rifampin once daily at least 1 hour before or 2 hours after the ingestion of food. On Day 22 (Cycle 2), participants were administered an oral dose of 600 mg of rifampin while in a fasted state in the clinic. Participants were then administered a single 3-hour IV infusion of ixabepilone 40 mg/m^2. On Days 23-28, participants self-administered a 600-mg oral dose of rifampin once daily at least 1 hour before or 2 hours after the ingestion of food. During Cycle 3 and beyond, participants received a single 3-hour IV infusion of ixabepilone at a dose of 40 mg/m^2 (unless their dose had been reduced) on Day 1 of each 21-day cycle for a maximum of 6 full cycles.
Period: Overall Study
Arm/Group | All Participants
Started | 15 (Number of participants treated)
Completed | 8
Not Completed | 7
Not completed — Study drug toxicity | 3
Not completed — Chest wall mass larger | 1
Not completed — Disease progression/relapse | 2
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (14)
Age, Customized [Number; unit: participants]
  < 65 years | 7
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 12
Race/Ethnicity, Customized [Number; unit: participants]
  White | 15
Race/Ethnicity, Customized [Number; unit: participants]
  Not Hispanic/Latino | 15
Body surface area (BSA) continuous [Mean (Standard Deviation); unit: square meter] — BSA is the measured or calculated surface of a human body.
  square meter | 1.9 (0.3)
Height continuous [Mean (Standard Deviation); unit: centimeter] | 173.5 (9.0)
Weight continuous [Mean (Standard Deviation); unit: kilogram] | 80.3 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax)
Description: Cmax was obtained directly from the concentration-time data.
Time Frame: Blood samples were collected on Day 1 (pre-dose, then 1h30, 3h, 3h15, 3h30, 4h, 6h and 8h), Day 2, Day 3, Day 4 and Day 8 during ixabepilone administration and repeated for Cycle 2 (Days 22-25 and 29) during ixabepilone and rifampin co-administration.
Population: Of the 15 patients in each group, only those with evaluable pharmacokinetic (PK) results are presented.
Measure: Geometric Mean (90% Confidence Interval); unit: nanogram (ng)/millilter(mL)
Groups:
- Ixabepilone: On Day 1 of Cycle 1, each participant received a single 3-hour IV infusion of ixabepilone 40 mg/m^2. (Participants then proceeded through the rest of Cycle 1 and on to further cycles - see the "ixabepilone + rifampin" treatment arm).
- Ixabepilone + Rifampin: Having already received ixabepilone on Day 1 of Cycle 1 (see the "ixabepilone" treatment arm), participants were administered an oral dose of 600 mg rifampin on in the clinic on Day 15. On Days 16-21, participants self-administered rifampin once daily, at least 1 hour before or 2 hours after the ingestion of food. On Day 22 (Cycle 2), participants were administered an oral dose of 600 mg of rifampin while in a fasted state in the clinic. Participants were then administered a single 3-hour IV infusion of ixabepilone 40 mg/m^2. On Days 23-28, participants self-administered a 600-mg oral dose of rifampin once daily at least 1 hour before or 2 hours after the ingestion of food. During Cycle 3 and beyond, participants received a single 3-hour IV infusion of ixabepilone at a dose of 40 mg/m^2 (unless their dose had been reduced) on Day 1 of each 21-day cycle for a maximum of 6 full cycles.
Arm/Group | Ixabepilone | Ixabepilone + Rifampin
Number analyzed (Participants) | 14 | 10
nanogram (ng)/millilter(mL) | 338.23 [281.78 to 405.99] | 308.37 [248.12 to 383.23]
Statistical Analysis 1: Comparison: Ixabepilone vs Ixabepilone + Rifampin; Two-way analyses of variance were performed on log-transformed values of Cmax. The factors in the analyses were participant and day. Point estimates and 90% confidence intervals for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale; Test type: Superiority or Other; Point estimate = 0.912, 90% CI 2-sided [0.751 to 1.106]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC [INF])
Description: AUC (INF) was obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: All treated participants who were evaluable for PK analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: nanogram (ng)*hour(hr)/mL
Arm/Group | Ixabepilone | Ixabepilone + Rifampin
Number analyzed (Participants) | 14 | 10
nanogram (ng)*hour(hr)/mL | 3028.70 [2425.48 to 3781.94] | 1713.07 [1473.74 to 1991.27]
Statistical Analysis 1: Comparison: Ixabepilone vs Ixabepilone + Rifampin; Two-way analyses of variance were performed on log-transformed values of (AUC [INF]). The factors in the analyses were participant and day. Point estimates and 90% confidence intervals for means and differences between means on the log scale were exponentiated to obtain estimates for geometric means and ratio of geometric means on the original scale; Test type: Superiority or Other; Point estimate = 0.566, 90% CI 2-sided [0.482 to 0.664]

3. Secondary Outcome: Number of Participants Who Died and Who Experienced Other Serious AEs (SAEs), Grade 3-4 AEs, Drug-related AEs and AEs Leading to Study Drug Discontinuation
Description: AEs:new untoward medical occurrences/worsening of pre-existing medical condition,whether or not related to study drug.SAE:AE resulting in death;life threatening;resulted in persistent/significant disability/incapacity;resulted in/prolonged existing hospitalization;a congenital anomaly/birth defect;overdose.Drug-related AEs: relationship to drug of certain;probable;possible;or missing.Participants who discontinued study due to AE were also recorded.AEs graded using National Cancer Institute (NCI) Common Toxicity Criteria (CTC),v3:Grade 1=mild,2=moderate, 3=severe,4=life threatening,5=death.
Time Frame: From Day 1 to 30 days after the last dose of study drug.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
participants
  Death | 0
  Other SAEs | 4
  Treatment-related AEs | 15
  Grade 3-4 AEs | 10
  Discontinuation due to AEs | 3

4. Secondary Outcome: Number of Participants With Grade 3-4 Hematology Abnormalities
Description: Abnormalities occurring at any time during the study were graded per NCI CTC, v3.0 criteria (Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening). Grade 3 and 4 criteria are given below. Neutrophils: Grade 3: 0.5 - <1.0x10^9/L, Grade 4: <0.5x10^9/L. Leukocytes: Grade 3: 1.0 - <2.0x10^9/L, Grade 4: <1.0x10^9/L. Neutrophils + bands (absolute): Grade 3: 0.5 - <1.0x10^9/L, Grade 4: <0.5x10^9/L. Hemoglobin: Grade 3:6.5 - <8.0g/dL, Grade 4: <6.5g/dL. Lymphocytes: Grade 3: 0.2 - <0.5x10^9/L, Grade 4: <0.2x10^9/L. Platelets: Grade 3: 25.0 - <50.0x10^9/L, Grade 4: <25.0x10.
Time Frame: Screening, Day 1, Day 8, Day 15, Day 22 and Day 29-36.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
participants
  Neutrophils (absolute) | 5
  Leukocytes | 6
  Neutrophils + bands (absolute) | 5
  Hemoglobin | 1
  Lymphocytes (absolute) | 6
  Platelet count | 0

5. Secondary Outcome: Number of Participants With Grade 3-4 Serum Chemistry Abnormalities in Alanine Aminotransferase, Aspartate Aminotransferase, Bilirubin, Albumin and Phosphorous
Description: Abnormalities occurring at any time during the study were graded per the NCI CTC (1=mild, 2=moderate, 3=severe, 4=life threatening). Grade 3 and 4 criteria were as follows: Alanine aminotransferase, aspartate aminotransferase and alkaline phosphatase: Grade 3: >5-20 x upper limit of normal (ULN), Grade 4: >20 x ULN. Bilirubin: Grade 3: >3-10 x ULN, Grade 4: >10 x ULN. Albumin: Grade 3: <2g/dL (Grade 4 not defined in NCI CTC). Creatinine: Grade 3: >3-6 x ULN, Grade 4: >6 x ULN. Phosphorous: Grade 3: 1-<2mg/dL, Grade 4: <1mg/dL.
Time Frame: Screening, Days 1 and 22.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
participants
  Alanine Aminotransferase | 0
  Aspartate Aminotransferase | 0
  Alkaline Phosphatase | 0
  Bilirubin | 0
  Albumin | 0
  Creatinine | 0
  Phosphorous (inorganic) | 1

6. Primary Outcome: Time Taken for Plasma Concentration to Reduce by 50 Percent or Apparent Terminal Plasma Elimination Half-life (T Half)
Description: T half was obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: All treated participants who were evaluable for PK analysis.
Measure: Mean (Standard Deviation); unit: Hrs
Arm/Group | Ixabepilone | Ixabepilone + Rifampin
Number analyzed (Participants) | 14 | 10
Hrs | 50.85 (18.59) | 36.45 (15.29)

7. Primary Outcome: Mean Residence Time Adjusted for Infusion Time (MRT [INF])
Description: (MRT [INF]) was obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: All treated participants who were evaluable for PK analysis.
Measure: Mean (Standard Deviation); unit: Hrs
Arm/Group | Ixabepilone | Ixabepilone + Rifampin
Number analyzed (Participants) | 14 | 10
Hrs | 50.93 (22.05) | 29.86 (15.31)

8. Primary Outcome: Total Body Clearance (CLT)
Description: CLT was obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: All treated participants who were evaluable for PK analysis.
Measure: Mean (Standard Deviation); unit: Litres(L)/hr
Arm/Group | Ixabepilone | Ixabepilone + Rifampin
Number analyzed (Participants) | 14 | 10
Litres(L)/hr | 28.36 (15.04) | 49.99 (17.19)

9. Primary Outcome: Volume of Distribution at Steady-state (Vss)
Description: Vss was obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: All treated participants who were evaluable for PK analysis.
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Ixabepilone | Ixabepilone + Rifampin
Number analyzed (Participants) | 14 | 10
L | 1323.26 (684.63) | 1447.54 (763.15)

10. Primary Outcome: Time to Reach Maximum Observed Concentration (T Max)
Description: T max was obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: All treated participants who were evaluable for PK analysis.
Measure: Median (Full Range); unit: Hrs
Arm/Group | Ixabepilone | Ixabepilone + Rifampin
Number analyzed (Participants) | 14 | 10
Hrs | 1.57 [1.5 to 3.3] | 1.50 [1.5 to 1.5]

11. Secondary Outcome: Number of Participants With Grade 3-4 Serum Chemistry Abnormalities in Calcium, Magnesium, Potassium, Sodium, Glucose and Uric Acid.
Description: Abnormalities occurring at any time during the study were graded per NCI CTC (1=mild, 2=moderate, 3=severe, 4=life threatening). Grade 3 and 4 criteria were as follows:Calcium: Grade 3: 6-<7 or >12.5-13.5mg/dL, Grade 4:<6 or >13.5mg/dL. Magnesium: Grade 3:0.6-<0.8 or >2.46-6.6mEq/L, Grade 4:<0.6 or >6.6mEq/L. Potassium: Grade 3:2.5-<3 or >6-7mmol/L, Grade 4:<2.5 or >7.0 mmol/L. Sodium: Grade 3:120-<130 or >155-160 mEq/L, Grade 4:<120 or >160mEq/L. Glucose: Grade 3:30-<40 or >250-500mg/dL, Grade 4:<30 or >500mg/dL. Uric acid: Grade 3:>ULN-10mg/dL with physiologic consequences, Grade 4:>10mg/dL.
Time Frame: Screening, Days 2 and 22.
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
Participants
  Calcium (total) | 0
  Magnesium (serum) | 0
  Potassium (serum) | 0
  Sodium (serum) | 1
  Glucose (serum) | 0
  Uric acid | 0

12. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Time of Last Quantifiable Concentration (AUC [0-T])
Description: AUC (0-T) was obtained directly from the concentration-time data.
Time Frame: as for outcome 1
Population: All treated participants who were evaluable for PK analysis.
Measure: Mean (Standard Deviation); unit: nanogram (ng)*hr/mL
Arm/Group | Ixabepilone | Ixabepilone + Rifampin
Number analyzed (Participants) | 14 | 10
nanogram (ng)*hr/mL | 3015.45 (1383.85) | 1478.31 (486.57)

13. Primary Outcome: Urine 6B-Hydroxycortisol to Cortisol Ratio on Day -1
Description: The urine 6B-hydroxycortisol to cortisol ratio is a measure of hepatic CYP3A4/3A5 activity, which is a potential marker of the rate of clearance of ixabepilone. The urine 6B-hydroxycortisol to cortisol ratios were calculated on Day -1.
Time Frame: Day -1 (0-8 hours and 8-24 hours), 24 hours before starting of ixabepilone administration.
Population: All treated participants who were evaluable for PK analysis.
Measure: Mean (Standard Deviation); unit: Ratio
Groups:
- All Participants: All participants who were enrolled into the study, 24 hours before ixabepilone administration on Day -1. Each participant received a single 3-hour IV infusion of ixabepilone 40 mg/m^2 on Day 1 of Cycle 1. Each participant was administered an oral dose of 600 mg of rifampin while in a fasted state on Day 22 (Cycle 2). Participants were then administered a single 3-hour IV infusion of ixabepilone 40 mg/m^2. On Days 23 through 28, participants self-administered a 600-mg oral dose of rifampin once daily at least 1 hour before or 2 hours after the ingestion of food during Cycle 2.
Arm/Group | All Participants
Number analyzed (Participants) | 14
Ratio
  0-8 hours | 10.04 (5.76)
  8-24 hours | 9.29 (5.84)

14. Secondary Outcome: Number of Participants With Clinically Meaningful Vital Signs Measures
Description: Vital signs were recorded throughout the study and included investigations related to body temperature, respiratory rate, seated blood pressure (systolic and diastolic), and heart rate. Normal ranges for the above are as follows: heart rate: 40 - 125 beats per minute (bpm); systolic BP: 65 - 200 millimeters of mercury (mmHg); diastolic BP: 40 - 120 mmHg; respiratory rate: 10 - 25 breaths per minute; temperature: 95 - 105F or 35 - 40.5C. The abnormalities displayed here are those considered "clinically significant" by the investigator and include abnormalities recorded at any time during study.
Time Frame: From screening to the off treatment visit.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
participants | 0

15. Primary Outcome: Urine 6B-Hydroxycortisol to Cortisol Ratio on Day 22
Description: as for outcome 13
Time Frame: Day 22 (0-8 hours and 8-24 hours) during ixabepilone and rifampin co-administration.
Population: All treated participants who were evaluable for PK analysis.
Measure: Median (Standard Deviation); unit: Ratio
Groups:
- Ixabepilone + Rifampin: Each participant was administered an oral dose of 600 mg of rifampin while in a fasted state on Day 22 (Cycle 2). Participants were then administered a single 3-hour IV infusion of ixabepilone 40 mg/m^2.
Arm/Group | Ixabepilone + Rifampin
Number analyzed (Participants) | 10
Ratio
  0-8 hours | 110.88 (101.91)
  8-24 hours | 62.42 (54.35)

16. Secondary Outcome: Number of Participants With Abnormal Physical Examination Findings
Description: Physical examination included height (screening only),weight,BSA,Eastern Cooperative Oncology Group Performance Status (ECOG PS),tendon reflexes,sensory function,motor strength. ECOG PS used to assess disease severity:score of 0 is fully active;1 is restricted physically strenuous activity;2 is ambulatory but unable to work;3 is capable of only limited self care;4 is completely disabled;5 is dead. Normal ranges:height:137-200cm or 54-79 inches;weight:40-135kg or 88-298 pounds (lbs);ECOG Scale:0-4. Abnormalities displayed here are those considered "clinically significant" by the investigator.
Time Frame: From screening to the off treatment visit.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
participants
  Weight-related abnormalities | 3
  Other physical examination abnormalities | 0

17. Secondary Outcome: QT Interval Corrected for Heart Rate (QTcF)
Description: QT interval corrected for heart rate (QTcF) was assessed using triplicate 12-lead serial electrocardiograms (ECGs) that were performed at selected times after the first dose of ixabepilone without rifampin and at matched times prior to the first dose of ixabepilone. Abnormalities occurring at any time during the study were recorded.
Time Frame: Data collected at 0, 1.5, 3, 4, 6, 8 and 24 hours after start of infusion.
Population: All participants treated with ixabepilone. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Mean (90% Confidence Interval); unit: millisecond
Groups:
- Ixabepilone: On Day 1 of Cycle 1, each participant received a single 3-hour IV infusion of ixabepilone 40 mg/m^2.
Arm/Group | Ixabepilone
Number analyzed (Participants) | 15
millisecond
  0 hour (n=9) | 3.44 [-2.06 to 8.95]
  1.5 hour (n=14) | 5.64 [0.54 to 10.74]
  3 hour (n=14) | 0.57 [-5.79 to 6.94]
  4 hour (n=11) | 7.82 [3.62 to 12.01]
  6 hour (n=13) | 6.54 [1.73 to 11.35]
  8 hour (n=3) | -10.70 [-31.61 to 10.28]
  24 hour (n=10) | -1.90 [-7.18 to 3.38]

18. Secondary Outcome: Number of Participants With Identified ECG Abnormalities
Description: Triplicate 12-lead serial ECGs were performed pre-dose (just prior to infusion), 1.5, 3 (just prior to end of the infusion even if infusion lasted for less than or more than planned 3 hrs), 4, 6, 8 and 24 hrs after start of ixabepilone infusion. Triplicate 12-lead serial ECGs were also to be performed on the date prior to dosing at times approximating post-dose schedule (pre-dose triplicate set of ECGs also qualified as the 24-hr baseline ECGs). Normal ranges for ECG are as follows: heart rate: 40 - 125 bpm; PR: 0.1 - 0.2 msec; QRS: 0.06 - 0.12 msec; QTC: 0.3 - 0.45 msec; QT: 0.3 - 0.5 msec.
Time Frame: Data collected at screening, Day -1 and Day 1 (at 0, 1.5, 3, 4, 6, 8 and 24 hours) after start of infusion.
Population: All participants treated with ixabepilone.
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 15
Participants
  Newly identified ECG abnormalities | 13
  Discontinuation due to ECG abnormalities | 1
  Abnormalities related to QT/QTc interval | 0
  Total number of ECG abnormalities | 13

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 4/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=15)
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 2
HYPERTENSION (Vascular disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
VOMITING (Gastrointestinal disorders) | 1
CHEST PAIN (General disorders) | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=15)
PHOTOPHOBIA (Eye disorders) | 1
LACRIMATION INCREASED (Eye disorders) | 1
HAEMOGLOBIN (Investigations) | 3
PLATELET COUNT (Investigations) | 1
NEUTROPHIL COUNT (Investigations) | 2
WEIGHT DECREASED (Investigations) | 3
HAEMOGLOBIN DECREASED (Investigations) | 3
WHITE BLOOD CELL COUNT (Investigations) | 1
PLATELET COUNT DECREASED (Investigations) | 3
NEUTROPHIL COUNT DECREASED (Investigations) | 2
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 4
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 1
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1
PALLOR (Vascular disorders) | 1
FLUSHING (Vascular disorders) | 1
HOT FLUSH (Vascular disorders) | 1
HYPOTENSION (Vascular disorders) | 1
ANXIETY (Psychiatric disorders) | 1
INSOMNIA (Psychiatric disorders) | 2
DEPRESSION (Psychiatric disorders) | 1
RESTLESSNESS (Psychiatric disorders) | 1
HEPATOMEGALY (Hepatobiliary disorders) | 1
HYPERSENSITIVITY (Immune system disorders) | 1
TREMOR (Nervous system disorders) | 2
HEADACHE (Nervous system disorders) | 3
AREFLEXIA (Nervous system disorders) | 1
DIZZINESS (Nervous system disorders) | 1
DYSGEUSIA (Nervous system disorders) | 6
PARAESTHESIA (Nervous system disorders) | 1
SENSORY DISTURBANCE (Nervous system disorders) | 1
NEUROPATHY PERIPHERAL (Nervous system disorders) | 4
RESTLESS LEGS SYNDROME (Nervous system disorders) | 1
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 3
NAUSEA (Gastrointestinal disorders) | 6
RETCHING (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 4
DIARRHOEA (Gastrointestinal disorders) | 8
DRY MOUTH (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 1
ORAL PAIN (Gastrointestinal disorders) | 1
STOMATITIS (Gastrointestinal disorders) | 2
CONSTIPATION (Gastrointestinal disorders) | 5
HAEMORRHOIDS (Gastrointestinal disorders) | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
RHINITIS (Infections and infestations) | 1
ORAL CANDIDIASIS (Infections and infestations) | 1
ANOREXIA (Metabolism and nutrition disorders) | 11
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 2
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 2
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 2
ANAEMIA (Blood and lymphatic system disorders) | 2
LYMPHOPENIA (Blood and lymphatic system disorders) | 2
NEUTROPENIA (Blood and lymphatic system disorders) | 2
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 1
RASH (Skin and subcutaneous tissue disorders) | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 9
PRURITUS (Skin and subcutaneous tissue disorders) | 2
URTICARIA (Skin and subcutaneous tissue disorders) | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 1
SKIN IRRITATION (Skin and subcutaneous tissue disorders) | 1
ADNEXA UTERI PAIN (Reproductive system and breast disorders) | 1
FALL (Injury, poisoning and procedural complications) | 1
EXCORIATION (Injury, poisoning and procedural complications) | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 7
LIMB DISCOMFORT (Musculoskeletal and connective tissue disorders) | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 4
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 1
PAIN (General disorders) | 1
CHILLS (General disorders) | 6
FATIGUE (General disorders) | 13
FEELING HOT (General disorders) | 3
EARLY SATIETY (General disorders) | 1
CHEST DISCOMFORT (General disorders) | 1
OEDEMA PERIPHERAL (General disorders) | 4
INFUSION SITE PAIN (General disorders) | 2
INFUSION SITE WARMTH (General disorders) | 1
MUCOSAL INFLAMMATION (General disorders) | 2
INJECTION SITE REACTION (General disorders) | 2
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.